CLINICAL TRIAL: NCT02133235
Title: The Need and the Effectiveness of Fiberoptic Bronchoscopy for Better Lung Collapse in Vedio-assisted Thoracic Operations Using Endobronchial Blockers
Brief Title: The Need of Fiberoptic Bronchoscopy for Placing an Endobronchial Blocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 201212175RINC
Record Dates: First submitted 2014-04-28; First posted 2014-05-07 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasms, Pulmonary; Thoracic Diseases
Keywords: endobronchial blocker; lung separation; vedio-assisted thoracic operation
MeSH Terms: conditions — Lung Neoplasms; Thoracic Diseases | interventions — Congresses as Topic; Auditory Perception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional (Active Comparator): insertion of endobronchial blocker and auscultation, fiberoptic confirmation and reposition
  Interventions: Procedure: conventional
- auscultation (Experimental): insertion endobronchial blocker by auscultation without conventional bronchoscopic reposition
  Interventions: Procedure: auscultation

INTERVENTIONS:
Procedure: conventional — insertion endobronchial blocker with the guidance of fiberoptic bronchoscopy
  Arms: conventional
Procedure: auscultation — insertion endobronchial blocker by auscultation, without the guidance of fiberoptic bronchoscopy
  Arms: auscultation

SUMMARY:
The need of fiberoptic bronchoscopy for placing an endobronchial blocker. Endobronchial blockers (EBB) have been presented effective and safe alternative for lung separation in vedio-assisted thoracoscopic (VATS) operations. In this study, the investigators will randomize the patients receiving VATS operation with EBB into two groups: one group will receive the conventional bronchoscopic guided EBBs placement, the other group receive two step procedure without confirmation by fiberoptic bronchoscopy.

DETAILED DESCRIPTION:
The need of fiberoptic bronchoscopy for placing an endobronchial blocker. Endobronchial blockers (EBB) have been presented effective and safe alternative for lung separation in vedio-assisted thoracoscopic (VATS) operations. However, there were previous reports showed that it takes longer time to position the EBB versus the double lumen tubes. Placing EBBs need three-step procedure (one is placing an endotracheal tube, the second is inserting the EBB, the third is confirmation of the position by fiberoptic bronchoscopy). In this study, the investigators will randomize the patients receiving VATS operation with EBB into two groups: one group will receive the conventional 3-step procedure, the other group receive two step procedure without confirmation by fiberoptic bronchoscopy.

ELIGIBILITY:
Inclusion criteria:

Lung separation by endobronchial blockers

Exclusion criteria:

Lung separation by conventional double lumen tube Lung separation with endobronchial blockers through

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Wang ML, Wang YP, Hung MH, Hsu HH, Chen JS, Yang FS, Cheng YJ. Is fibre-optic bronchoscopy necessary to confirm the position of rigid-angled endobronchial blockers before thoracic surgery? A randomized controlled trial. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):241-246. doi: 10.1093/ejcts/ezx260. PMID 28950380

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Fiberoptic Brochoscopy Group: patients receiving VATS operations with endobronchial blockers with procedures: endotracheal intubation, insertion of endobronchial blocker and auscultation, fiberoptic confirmation and reposition
- Auscultation Group: patients receiving vedio-assisted thoracic operations by endobronchial blocker with procedures: endotracheal intubation, insertion endobronchial blocker with auscultation without conventional bronchoscopic reposition
Period: Overall Study
Arm/Group | Conventional Fiberoptic Brochoscopy Group | Auscultation Group
Started | 55 | 57
Completed | 55 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auscultation Group | Conventional Fiberoptic Brochoscopy Group | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 40 | 83
  >=65 years | 14 | 15 | 29
Age, Continuous [Mean (Full Range); unit: years] | 58 [30 to 79] | 58 [35 to 79] | 58 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 20 | 50
  Male | 27 | 35 | 62
Region of Enrollment [Number; unit: participants]
  Taiwan | 57 | 55 | 112

OUTCOME MEASURES:

1. Primary Outcome: Surgical Grading for Lung Isolation
Description: A: Optimal; B: Lung distension; C: Poor endobronchial blocker placement
Time Frame: 10-15 minutes
Measure: Number; unit: participants
Groups:
- Left-sided VATS, Auscultation Group: patients receiving left-sided vedio-assisted thoracic operations by endobronchial blocker with procedures: endotracheal intubation, insertion of endobronchial blocker, confirmation of endobronchial blocker position by auscultation only
- Left-sided VATS, Conventional Fiberoptic Brochoscopy Group: patients receiving left-sided VATS operations with endobronchial blockers with procedures: endotracheal intubation, insertion of endobronchial blocker, confirmation of endobronchial blocker position by conventional fiberoptic brochoscopy group
- Right-sided VATS, Auscultation Group: patients receiving right-sided vedio-assisted thoracic operations by endobronchial blocker with procedures: endotracheal intubation, insertion of endobronchial blocker, confirmation of endobronchial blocker position by auscultation only
- Right-sided VATS, Conventional Fiberoptic Bronchoscopy Group: patients receiving right-sided VATS operations with endobronchial blockers with procedures: endotracheal intubation, insertion of endobronchial blocker, confirmation of endobronchial blocker position by conventional fiberoptic brochoscopy group
Arm/Group | Left-sided VATS, Auscultation Group | Left-sided VATS, Conventional Fiberoptic Brochoscopy Group | Right-sided VATS, Auscultation Group | Right-sided VATS, Conventional Fiberoptic Bronchoscopy Group
Number analyzed (Participants) | 22 | 28 | 32 | 30
participants
  A: Optimal | 12 | 13 | 15 | 14
  B: Lung distension | 10 | 11 | 13 | 12
  C: Poor endobronchial blocker placement | 0 | 4 | 4 | 4

2. Primary Outcome: Time Required for Proper Placement of the Endobronchial Blocker
Time Frame: 10-15 minutes
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Left-sided VATS, Auscultation Group: patients receiving left-sided vedio-assisted thoracic operations by endobronchial blocker with procedures: endotracheal intubation, insertion endobronchial blocker with auscultation without conventional bronchoscopic reposition
- Left-sided VATS, Conventional Fiberoptic Brochoscopy Group: patients receiving left-sided VATS operations with endobronchial blockers with procedures: endotracheal intubation, insertion of endobronchial blocker and auscultation, fiberoptic confirmation and reposition
- Right-sided VATS, Auscultation Group: patients receiving right-sided vedio-assisted thoracic operations by endobronchial blocker with procedures: endotracheal intubation, insertion endobronchial blocker with auscultation without conventional bronchoscopic reposition
- Right-sided VATS, Conventional Fiberoptic Bronchoscopy Group: patients receiving right-sided VATS operations with endobronchial blockers with procedures: endotracheal intubation, insertion of endobronchial blocker and auscultation, fiberoptic confirmation and reposition
Arm/Group | Left-sided VATS, Auscultation Group | Left-sided VATS, Conventional Fiberoptic Brochoscopy Group | Right-sided VATS, Auscultation Group | Right-sided VATS, Conventional Fiberoptic Bronchoscopy Group
Number analyzed (Participants) | 25 | 25 | 32 | 30
seconds | 138.5 (25.5) | 130 (20) | 89.6 (9.3) | 141.1 (16.4)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Conventional Fiberoptic Brochoscopy Group | Auscultation Group
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/57
Other Adverse Events (participants affected / at risk) | 0/55 | 3/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Fiberoptic Brochoscopy Group (N=55) | Auscultation Group (N=57)
Failure for optimal lung isolation (Surgical and medical procedures) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No